CLINICAL TRIAL: NCT06946264
Title: Characterization of Bronchodilator Response in Children With Bronchiolitis Using Phenotypic and Genotypic Features
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Andrea Rivera-Sepulveda, Associate Professor, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1866573
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Bronchiolitis; Bronchodilator Agents
Keywords: double-blind randomized clinical trial
MeSH Terms: conditions — Bronchiolitis | interventions — Albuterol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bronchodilator arm (Experimental): Children with bronchiolitis will be randomized to an intervention arm to be administered as a nebulization (albuterol sulfate 2.5mg/ 3mL inhalation solution). The intervention drug will be placed in a sealed manila envelope, randomized in advance by a Nemours Investigational Drug Pharmacist, and stored in the ED pyxis.
  Interventions: Drug: Albuterol Sulfate, 2.5 Mg/3 mL (0.083%) Inhalation Solution
- Normal saline arm (Placebo Comparator): Children with bronchiolitis will be randomized to an intervention arm to be administered as a nebulization (sodium chloride 0.9%/ 3mL inhalation solution). The intervention drug will be placed in a sealed manila envelope, randomized in advance by a Nemours Investigational Drug Pharmacist, and stored in the ED pyxis.
  Interventions: Drug: Sodium Chloride 0.9% Inhl 3Ml

INTERVENTIONS:
Drug: Albuterol Sulfate, 2.5 Mg/3 mL (0.083%) Inhalation Solution — Children with bronchiolitis will be randomized to an intervention arm to be administered as a nebulization (albuterol sulfate 2.5mg/ 3mL inhalation solution). The intervention drug will be placed in a sealed manila envelope, randomized in advance by a Nemours Investigational Drug Pharmacist, and stored in the ED pyxis.
  Arms: Bronchodilator arm
Drug: Sodium Chloride 0.9% Inhl 3Ml — Children with bronchiolitis will be randomized to an intervention arm to be administered as a nebulization (sodium chloride 0.9% 3mL inhalation solution). The intervention drug will be placed in a sealed manila envelope, randomized in advance by a Nemours Investigational Drug Pharmacist, and stored in the ED pyxis.
  Arms: Normal saline arm

SUMMARY:
Bronchiolitis is the leading cause of pediatric morbidity and healthcare costs. Despite the commonplace use of bronchodilator treatments, like albuterol, in conditions like asthma, their efficacy in bronchiolitis remains controversial due to the heterogeneity in patient response. Although studies indicate that bronchodilators do not enhance outcomes in bronchiolitis, meta-analyses can obscure the heterogeneity of treatment effects. While bronchodilator response genetics have not been explored in bronchiolitis, treatment effectiveness variations often depend on genomic factors. Genome-wide association studies (GWAS) have linked genetic variants with bronchodilator response and outcomes in childhood asthma, suggesting a bronchodilator-responsive genotype. This proposal aims to extend this paradigm to bronchiolitis, addressing the gap in knowledge where GWAS and clinical characteristics intersect. The proposed study's objective is to characterize phenotypic and genotypic variations of children with bronchiolitis and their association with bronchodilator response. We hypothesize that children with bronchiolitis who exhibit clinical and historical characteristics associated with atopy and specific physical findings have genetic variants linked to bronchodilator response. To achieve this, we propose to (Aim 1) define airway responsiveness to bronchodilator treatment in children with bronchiolitis using the change in respiratory score, (Aim 2a) identify the associations between candidate genetic variants and bronchodilator response among children with bronchiolitis, and (Aim 2b) determine the associations between candidate genetic variants and clinical patient data to identify bronchodilator-responsive children with bronchiolitis. A prospective, double-blind, randomized, placebo-controlled trial of a single albuterol dose in children aged 3 to 24 months presenting with bronchiolitis to the emergency department will be conducted to achieve these aims. Patient information and respiratory assessment outcomes will be collected before and after intervention. Blood, urine, DNA buccal swabs, and nasopharyngeal swabs will also be collected. Completion of these aims will result in a novel clinical prediction model for bronchodilator response determination in bronchiolitis, integrating clinical, physical, and genetic data. Furthermore, this research supports the candidates' career development goals of advancing training in clinical trial research design and execution and becoming an expert in clinical and translational methods to enhance pediatric emergency department health and outcomes. Ultimately, this work will inform an R01 application to validate an evidence-based prediction rule for identifying bronchodilator-responsive children with bronchiolitis through a multi-center emergency medicine research network, optimizing therapeutic approaches, and reducing resource use in those with a low likelihood of bronchodilator response.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 to 24 months of age
* Clinical diagnosis of bronchiolitis by the treating provider(s), defined by the American Academy of Pediatrics as a clinical syndrome involving lower respiratory tract symptoms
* Children who either have no history of prematurity or have a history of prematurity but without associated co-morbidities
* Emergency department (ED) visit to seek care at Nemours Children's Health-Florida (NCH-FL)

Exclusion Criteria:

* Patients previously enrolled in the PI's K12 study
* Documented history of asthma or reactive airway disease
* Co-morbidities affecting airway response (e.g., chronic lung disease, bronchopulmonary dysplasia, bronchiectasis, congenital heart disease, immunodeficiency, neurologic condition)
* Diagnosis of pneumonia by chest radiography
* Inhaled, nebulized, or oral corticosteroid use within 72 hours of ED evaluation
* Inhaled, nebulized, or oral bronchodilator administration within 4 hours of ED arrival

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimum Clinically Important Difference (Aim 1) | Immediately after the intervention
  Identify the minimum clinically important difference (MCID) in the modified Tal score (MTS) in children with bronchiolitis from parents/ caregivers and treating providers' perceived improvement in respiratory response. The minimum clinically important difference (MCID) is a 15-point scale, ranging from -7 (very much worse) to +7 (very much improved), as assessed by responses from the caregiver(s) and the treating provider(s). A response of +1 to +2 will be interpreted as a "small" perceived improvement in respiratory function.
  The modified Tal score (MTS) includes respiratory parameters documented as part of the ED standard of care. The MTS score ranges from 0 to 12 points, with higher scores indicating greater respiratory distress.
Candidate genetic variants (Aim 2) | through study completion, an average of 1 year
  Identify candidate single nucleotide polymorphisms (SNPs), rank-ordered by the strength of their association with the modified Tal score (delta) respiratory score based on an odds ratio (dichotomous response) or a beta coefficient (continuous response) and filtered by adjusted p-value.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical data that will be preserved and shared are demographical data, history of prematurity, immunizations, history of corticosteroid use, past medical history, family history, environmental exposure, pulmonary history, randomized drug administered, and physical exam data, among other data pertinent to the study. Clinical data from data collection forms will be preserved and shared. Genomic data that will be preserved and shared will include variant calls from genotyping microarrays with imputation. Clinical data sets will be submitted to the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) in .CSV format. Genomic data sets will be submitted to the Database of Genotypes and Phenotypes (dbGaP, NCBI, NIH) in CRAM, and VCF format.
Supporting Information: CSR
Time Frame: The repository will make the data accessible within 2 years of the last patient's enrollment or no later than the date of publication, whichever is sooner.

REFERENCES:
- [Background] McCulloh RJ, Smitherman SE, Koehn KL, Alverson BK. Assessing the impact of national guidelines on the management of children hospitalized for acute bronchiolitis. Pediatr Pulmonol. 2014 Jul;49(7):688-94. doi: 10.1002/ppul.22835. Epub 2013 Jul 19. PMID 23868897
- [Background] Knapp JF, Simon SD, Sharma V. Variation and trends in ED use of radiographs for asthma, bronchiolitis, and croup in children. Pediatrics. 2013 Aug;132(2):245-52. doi: 10.1542/peds.2012-2830. Epub 2013 Jul 22. PMID 23878045
- [Background] Willson DF, Horn SD, Hendley JO, Smout R, Gassaway J. Effect of practice variation on resource utilization in infants hospitalized for viral lower respiratory illness. Pediatrics. 2001 Oct;108(4):851-5. doi: 10.1542/peds.108.4.851. PMID 11581435
- [Background] Gong C, Byczkowski T, McAneney C, Goyal MK, Florin TA. Emergency Department Management of Bronchiolitis in the United States. Pediatr Emerg Care. 2019 May;35(5):323-329. doi: 10.1097/PEC.0000000000001145. PMID 28441240
- [Background] Viswanathan M, King VJ, Bordley C, Honeycutt AA, Wittenborn J, Jackman AM, Sutton SF, Lohr KN. Management of bronchiolitis in infants and children. Evid Rep Technol Assess (Summ). 2003 Jan;(69):1-5. No abstract available. PMID 12624885
- [Background] Gadomski AM, Scribani MB. Bronchodilators for bronchiolitis. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD001266. doi: 10.1002/14651858.CD001266.pub4. PMID 24937099
- [Background] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312
- [Background] Pelletier AJ, Mansbach JM, Camargo CA Jr. Direct medical costs of bronchiolitis hospitalizations in the United States. Pediatrics. 2006 Dec;118(6):2418-23. doi: 10.1542/peds.2006-1193. PMID 17142527
- [Background] Hasegawa K, Tsugawa Y, Brown DF, Mansbach JM, Camargo CA Jr. Trends in bronchiolitis hospitalizations in the United States, 2000-2009. Pediatrics. 2013 Jul;132(1):28-36. doi: 10.1542/peds.2012-3877. Epub 2013 Jun 3. PMID 23733801
- [Background] Willer RJ, Coon ER, Harrison WN, Ralston SL. Trends in Hospital Costs and Levels of Services Provided for Children With Bronchiolitis Treated in Children's Hospitals. JAMA Netw Open. 2021 Oct 1;4(10):e2129920. doi: 10.1001/jamanetworkopen.2021.29920. PMID 34698848
- [Background] Keren R, Luan X, Localio R, Hall M, McLeod L, Dai D, Srivastava R; Pediatric Research in Inpatient Settings (PRIS) Network. Prioritization of comparative effectiveness research topics in hospital pediatrics. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1155-64. doi: 10.1001/archpediatrics.2012.1266. PMID 23027409
- [Background] Meissner HC. Viral Bronchiolitis in Children. N Engl J Med. 2016 Jan 7;374(1):62-72. doi: 10.1056/NEJMra1413456. No abstract available. PMID 26735994
- [Background] Fujiogi M, Goto T, Yasunaga H, Fujishiro J, Mansbach JM, Camargo CA Jr, Hasegawa K. Trends in Bronchiolitis Hospitalizations in the United States: 2000-2016. Pediatrics. 2019 Dec;144(6):e20192614. doi: 10.1542/peds.2019-2614. Epub 2019 Nov 7. PMID 31699829

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT06946264/Prot_SAP_000.pdf